CLINICAL TRIAL: NCT04774757
Title: Curative Systemic Therapy Sequenced Radical Surgery for Synchronous Isolated Paraaortic Lymph Node Metastasis of Colorectal Cancer
Brief Title: Systemic Therapy Sequenced Isolated PALND for mCRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Guosheng Wu, Chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Synchronous isolated PALND
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Synchronous Isolated Para-aortic Lymph Node Metastasis; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic therapy sequenced PALND (Experimental): All received systemtic therapy (at most two lines).
  Interventions: Procedure: Para-aortic lymph node dissection

INTERVENTIONS:
Procedure: Para-aortic lymph node dissection — Para-aortic lymph node dissection was defined as the dissection of para-aortic lymph nodes located below renal vein and above the bifurcation of iliac artery.

SUMMARY:
The study aims to estimate the efficacy and safety of systemic therapy sequenced radical surgery in treating patients with synchronous isolated para-aortic lymph node metastasis of colorectal cancer.

DETAILED DESCRIPTION:
Patients with synchrnous isolated para-aortic lymph node metastasis of colorectal cancer receiving systemtic therapy (at most two lines), radiologically assessed efficacious, and assessed by MDT that are potential to reach no evidence of disease (NED) were included in our trial. All included patients receive para-aortic lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment is >= 18 and <= 75 years
2. ECOG PS 0-1
3. Histologically confirmed colorectal carcinoma
4. Synchronous metastatic colorectal cancer with isolated para-aortic lymph node metastases: In the preoperative examination of positron emission tomography CT and abdominopelvic CT, metastasis was noted when the diameter of the PALN was 10 mm or greater and had irregular shape.
5. Single-organ para-aortic lymph node metastasis (PLANM) who are potential to receive surgery and achieve no evidence of disease (NED).
6. Adequate liver, renal and bona marrow function.
7. Signing written informed consent

Exclusion Criteria:

1. In addition to PALN metastasis, distant metastases such as lung, liver, peritoneum and bone were presen and in instances when the renal vein was in the upward spread path of the LN metastasis.
2. Unable to achieve NED
3. Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention, Or a history of myocardial infarction in the last 12 months.
4. Those with other history of malignant disease in the last 5 years, except for cured skin cancer and cervical carcinoma in situ.
5. Organ transplantation requires immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year DFS | From date of recruiment until the date of disease recurrece, assessed up to 3 years
  Time with no recurrence of the diseases.

SECONDARY OUTCOMES:
5-year OS | Up to 5 years
  From date of recruitment until the date of death from any cause, assessed up to 5 years.
LFS | From date of recruiment until the date of paraaortic lymph node recurrece, assessed up to 5 years
  Time with no recurrence of the paraaortic lymph node region.
1-year DFS | From date of recruiment until the date of disease recurrece, assessed up to 1 years
  Time with no recurrence of the diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No